CLINICAL TRIAL: NCT01412632
Title: Deep Sedation in Spontaneously Breathing Patients Combined With Local Anesthesia Versus General Anesthesia in Gynecological Patients at Same Day Surgical at Hospitalsenheden Horsens
Brief Title: Comparing Two Types of Sedation to Gynaecological Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Horsens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010-023843-13
Record Dates: First submitted 2011-06-15; First posted 2011-08-09 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2013-08

CONDITIONS: Transcervical Resection of Endometrium; Transcervical Resection of Fibroids; Transcervical Resection of Polyp
MeSH Terms: interventions — Remifentanil; Propofol; Prilocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- General vs deep sedation (Experimental): General anesthesia: remifentanil and propofol Deep sedation: remifentanil, propofol and citanest
  Interventions: Drug: Remifentanil, propofol and citanest

INTERVENTIONS:
Drug: Remifentanil, propofol and citanest — iv remifentanil iv propofol im citanest

SUMMARY:
The primary endpoint is to investigate the difference in pain between patients who receive deep sedation with spontaneous breathing versus patients who receive general anesthesia.

DETAILED DESCRIPTION:
Investigate the difference between two types of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* females
* are having a TCRE, TCRF or TCRP
* speak and understand Danish
* no mental problems

Exclusion Criteria:

* <18 years old
* don´t speak or understand Danish
* mental problems
* Lung problems
* BMI >40
* Big fibroma: >3x3 cm
* abuser
* Allergy towards i Propofol, Remifentanil and/or Citanest
* pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
pain on a NRS-scale from 0 to 10 | up to 14 days
  Measuring postoperative pain in TCRE, TCRF or TCRP patients

SECONDARY OUTCOMES:
PONV | postoperative and 2 weeks after discharge
Time | 1 day
  Operating time Recovery time Discharge time
Medicin | 1 day
  The type and quantity of painkillers and nausea medication. Remifentanil, propofol, citanest, efedrin og atropin.
After discharge outcome measures | 2 weeks
  Previous anestetics, pain, PONV, fever, bleeding, discharge time.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Filipovski, Principal Investigator — Regionshospital Horsens
Locations (1):
- Regionshospitalet Horsens, Horsens, Region Midt, Denmark